CLINICAL TRIAL: NCT04796857
Title: Tislelizumab in Combination With Lenalidomide in in Patients With Relapsed or Refractory Elderly Patients With Non-GCB Diffuse Large B Cell Lymphoma: a Prospective Phase Ib/II, Multicentre, Open-label, Single-arm Trial
Brief Title: Tislelizumab in Combination With Lenalidomide in Refractory and Relapsed Elderly Patients With Non-GCB DLBCL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huiqiang Huang (Other)
Responsible Party: Sponsor-Investigator, Huiqiang Huang, professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TALEND
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Non-GCB/ABC Diffuse Large B-Cell Lymphoma; High-grade B-cell Lymphoma; Follicular Lymphoma Grade IIIb; Transformed Lymphoma; EBV-Positive DLBCL, Nos; ALK-Positive Anaplastic Large Cell Lymphoma
Keywords: DLBCL; Non-GCB/ABC; Relapsed; Refractory; Elderly Patients
MeSH Terms: conditions — Pyloric Stenosis, Hypertrophic; Recurrence | interventions — spartalizumab; tislelizumab; Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab in Combination With Lenalidomide (Experimental): On the day of tislelizumab infusion, lenalidomide should be taken 30 minutes after the end of tislelizumab infusion
  Interventions: Drug: PD-1 Antibody; Drug: Lenalidomide

INTERVENTIONS:
Drug: PD-1 Antibody — Tislelizumab will be administered every 4 weeks up to 6 cycles during induction phase if patients get CR or PR after induction phase.
  Other Names: Tislelizumab
Drug: Lenalidomide — Phase I: dose escalation phase. Patients will oral dosage as 10mg, 20mg, per day. Aim to evaluate MTD and DLT, RP2D.
  Phase II：Patients continuous oral lenalidomide as RP2D up to 6 cycles during induction phase
  Other Names: revlimid

SUMMARY:
Aim of this study will evaluate the efficacy and safety of tislelizumab in combination with lenalidomide in in patients with relapsed or refractory Elderly Patients with non-GCB Diffuse Large B Cell Lymphoma

DETAILED DESCRIPTION:
Elderly patients with relapsed /refractory non-GCB diffuse large B cell lymphoma usually have a bad prognosis. These patients cannot be treated successfully or tolerated the conventional chemotherapy. Lenalidomide has a unique therapeutic effect in Non-GCB DLBCL. Some studies have shown that the combination of lenalidomide and PD-1 antibody shows a synergistic effect in the exploration of DLBCL, and the patients are well tolerated.The investigators will evaluate the efficacy and safety of tislelizumab in combination with lenalidomide in the elderly patients with relapsed refractory non-GCB DLBCL failed from second line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers who signed informed consent.
2. Age range 60-75 years old; male or female
3. DLBCL, or follicular lymphoma grade 3B, or transformed DLBCL, EBV (+) DLBCL, ALK (+) DLBCL, high-grade lymphoma were confirmed by histopathology examination;
4. Failed from standard first-line rituximab-contained chemotherapy, and relapsed or refractory after second-line regimens with or without rituximab.
5. ECOG performance status 0-1.
6. Estimated survival time > 3 months.
7. There must be at least one evaluate able or measurable lesion that meets the LYRIC 2016 Malignant Lymphoma criteria [evaluable lesion: 18F-fluorodeoxyglucose/Positron Emission Tomography (18FDG/PET) examination showing increased lymph node or extranodal uptake (higher than liver) and PET and/or computed tomography (Computed Tomography) CT) features are consistent with lymphoma findings; lesions can be measured: nodular lesions > 15mm or extranodal lesions > 10mm (if the only measurable lesion has received radiotherapy in the past, there must be evidence of radiological progress after radiotherapy), and accompanied by increased 18FDG uptake). Except for this, there is no measurable increase in diffuse 18FDG uptake in the liver;
8. Adequate organ and bone marrow function, no severe hematopoietic dysfunction, cardiac, pulmonary, liver, kidney, thyroid dysfunction and immune deficiency (no blood transfusion, granulocyte colony stimulating factor or other medical support was received within 14 days prior to the use of the research drug): 1) The absolute value of neutrophils (>1.5×10^9/L); 2) platelet count (> 75×10^9/L); 3) Hemoglobin (> 9 g/dL); 4) Upper Limit Normal (ULN) or creatinine clearance rate (>40 mL/min) of serum creatinine (<1.5 times normal value upper limit) (estimated by Cockcroft-Gault formula); 5) Serum total bilirubin < 1.5 times ULN; 6) Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) = 2.5 times ULN; 7) Prior chemotherapy and radiotherapy should have been completed more than 4 weeks. Coagulation function: International Normalized Ratio (INR) = 1.5 times ULN; Prothrombin Time (PT), Activated Partial Thromboplastin Time (APTT) = 1.5 times ULN (unless the subject is receiving anticoagulant therapy and PT and APTT are using anticoagulant therapy at screening time). Within the expected range; 8) Thyrotropin (TSH) or free thyroxine (FT4) or free triiodothyronine (FT3) were all within the normal range (+10%);
9. There was no evidence that subjects had difficulty breathing at rest, and the measured value of pulse oximetry at rest was more than 92%;
10. Participants must pass a pulmonary function test (PFT) to confirm that forced expiratory volume (FEV1)/forced vital capacity (FVC) in the first second is more than 60%, unless it is a large mediastinal mass caused by lymphoma that cannot meet this standard; carbon monoxide diffusion (DLCO), FEV1 and FVC are all above 50% of the predicted value; all PFT results must be obtained within four weeks before the first administration;
11. Female patients of childbearing age must have a negative pregnancy test at the time of enrollment and are willing to use reliable contraceptive methods, i.e. barrier methods, oral contraceptives, implant methods, skin contraception, long-acting injection contraceptives, intrauterine devices, or tubal ligation;
12. Paraffin tissue specimens or fresh puncture tissue specimens are available.

Exclusion Criteria:

1. Hemophagocytic syndrome;
2. Primary central nervous system lymphoma or secondary central nervous system involvement;
3. Received allogeneic organ transplantation in the past;
4. The study began with Allo-HSCT(Allogeneic Hematopoietic Stem Cell Transplantation) within 3 years before treatment;
5. Participating in other clinical studies, or less than 4 weeks from the end of the previous clinical study;
6. Accepted autologous hemopoietic stem cell transplantation within 3 month before treatment;
7. Previously treated with lenanlidomde or immune checkpoint inhibitors within 1 year;
8. Thalidomide intolerance;
9. Peripheral neurotoxicity > grade 1;
10. Under risk of thromboembolism and are unwilling to prevent venous thromboembolism;
11. Patients with active autoimmune diseases requiring systematic treatment in the past two years (hormone replacement therapy is not considered systematic treatment, such as type I diabetes mellitus, hypothyroidism requiring only thyroxine replacement therapy, adrenocortical dysfunction or pituitary dysfunction requiring only physiological doses of glucocorticoid replacement therapy); Patients with autoimmune diseases who do not require systematic treatment within two years can be enrolled;
12. Begin the study on subjects requiring systemic glucocorticoid therapy or other immunosuppressive therapy for a given condition within 14 days before treatment [allowing subjects to use local, ocular, intra-articular, intranasal and inhaled glucocorticoid therapy (with very low systemic absorption); and allowing short-term (< 7 days) glucocorticoid prophylaxis (e.g., contrast agent overdose) Sensitivity) or for the treatment of non-autoimmune diseases (e.g. delayed hypersensitivity caused by contact allergens), except for tumor reduction due to large tumor burden (prednisone 30mg, bid × 5 days or equivalent dose of other glucocorticoid therapy);
13. In the past five years, patients with other malignant tumors have undergone radical treatment, except for basal cell carcinoma of skin, squamous cell carcinoma of skin, carcinoma in situ of breast and carcinoma in situ of cervix;
14. Begin the study and receive systemic antineoplastic therapy within 28 days before treatment, including chemotherapy, immunotherapy, biotherapy (cancer vaccine, cytokines, or growth factors that control cancer), etc.;
15. The study began with major surgery within 28 days before treatment or radiotherapy within 90 days before treatment;
16. Start the study and receive Chinese herbal medicine or Chinese 12.patent medicine treatment within 7 days before treatment;
17. Begin research on live vaccination (except influenza attenuated vaccine) within 28 days before treatment;
18. History of human immunodeficiency virus (HIV) infection and/or patients with acquired immunodeficiency syndrome are known;
19. Patients with active hepatitis B or active hepatitis C. Patients who are positive for hepatitis B Surface Antigen (HBsAg) or hepatitis C Virus (HCV) antibodies at screening stage must pass further detection of hepatitis B Virus (HBV) DNA titer (no more than 2500 copies/mL or 500 IU/mL) and HCV RNA (no more than the lower limit of the detection method) in the row. In addition to active hepatitis B or hepatitis C infections requiring treatment, group trials can be conducted. Hepatitis B carriers, stable hepatitis B (DNA titer should not be higher than 2500 copies/mL or 500 IU/mL) after drug treatment, and cured hepatitis C patients can be enrolled in the group;
20. Patients with active pulmonary tuberculosis;
21. Start studying any active infections requiring systemic anti-infective treatment within 14 days of treatment.
22. Pregnant or lactating women;
23. People with known history of alcoholism or drug abuse;
24. History of interstitial lung disease or non-infectious pneumonia.
25. Subjects who had previously had non-infectious pneumonia caused by drugs or radiation but had no symptoms were allowed to enter the group;
26. QTCF interval > 450 msec;
27. Past psychiatric history; incapacitated or restricted;
28. According to the researchers' judgment, patients' underlying condition may increase their risk of receiving research drug treatment, or confuse their judgment on toxic reactions;
29. Other researchers consider it unsuitable for patients to participate in this study.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-31 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR), Investigator-Assessed | up to 24 months
  Overall response was determined on the basis of investigator assessments according to lymphoma response to immunomodulatory therapy criteria (LYRIC) for Malignant Lymphoma, 2016. Tumor assessments were performed with CT/MRI with or without PET.
The optimal dosage of lenalidomide | up to 6 months
  Maximum tolerable dose（MTD）and dose-limiting toxicity（DLT）of lenalidomide will be conducted in Phase Ib clinical studies. MTD and DLT is defined as protocol-defined lenalidomide related events.

SECONDARY OUTCOMES:
Progression-free Survival | Time Frame: up to 36 months
  The time between the start of randomization and the progression of the tumor (any aspect) or (for any reason) death
Overall Survival | up to 36 months
  Time from randomization to death for any reason Time from randomization to death for any reason Time from randomization to death for any reason Time from randomization to death for any reason
Duration of Response | Time Frame: up to 36 months
  The time from the first assessment of CR or PR to PD (progressive disease) or death from any cause
Time To Progression | up to 36 months
  Time from randomization to PD
Percentage of Participants With Adverse Events (AEs) | Up to 36 months
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Huiqiang Huang, Professor, Principal Investigator — huanghq@sysucc.org.cn
Locations (1):
- Department of Medical Oncology, Sun Yat-sen University Cancer Center,, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No